CLINICAL TRIAL: NCT03543241
Title: MyoStrain CMR Testing of Ischemia With Low Levels of Stress
Status: Completed | Type: Observational
Sponsor: Myocardial Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: VAL-1006P(A)
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Myocardial Dysfunction
Keywords: Strain
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- MyoStrain: Patients with suspected CAD and scheduled for cardiac catheterization will receive traditional CMR wall motion stress testing with MyoStrain software analysis of myocardial ischemia and viability.
  Interventions: Diagnostic Test: MyoStrain

INTERVENTIONS:
Diagnostic Test: MyoStrain — Prior to cardiac catheterization, patients will be stress testing with low dose Dobutamine to evaluate wall motion, segmental, and global myocardial strain at rest and under stress to determine the accuracy of detecting ischemia and viability of myocardial tissue.

SUMMARY:
This prospective, observational study evaluates the accuracy of stress testing with the MyoStrain SENC CMR Imaging System to detect myocardial ischemia and viability in patients with suspected coronary artery disease using low levels of stress.

DETAILED DESCRIPTION:
This prospective, single center study evaluates the MyoStrain SENC CMR Imaging System for the detection of myocardial ischemia and viability during conventional Cardiac Magnetic Resonance (CMR) wall motion stress testing. Patients with known or suspected coronary artery disease and scheduled for cardiac catheterization will be consented for inclusion in the study and evaluated during stress testing with low dose Dobutamine as the stressor agent. Data obtained with the MyoStrain SENC CMR Imaging System will be for observational purposes and will not be used to alter patient management.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected Coronary Artery Disease
* Symptoms potentially due to CAD; stable angina
* Positive imaging stress test or negative stress test but typical angina or anginal equivalent
* Negative Troponin with unstable angina
* Invasive coronary angiography planned within 3 months of CMR
* Provided written consent

Exclusion Criteria:

* Pregnancy
* Contraindication to Magnetic Resonance Imaging
* Prior allergy to Dobutamine
* Severe aortic stenosis
* Hypertrophic Cardiomyopathy
* Clinically significant Ventricular Tachycardia that would prohibit Dobutamine administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected coronary artery disease scheduled for cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Ischemic CAD Detection | Up to coronary angiography within 1 month of standard CMR stress testing
  Sensitivity of correctly identifying ischemic coronary artery disease based on cardiac catheterization results using low dose Dobutamine stress testing with MyoStrain software

SECONDARY OUTCOMES:
Specificity of Ischemic CAD Detection | Up to coronary angiography within 1 month of standard CMR stress testing
  Specificity of correctly screening patients with ischemic coronary artery disease based on cardiac catheterization results using MyoStrain stress testing with low dose Dobutamine

CONTACTS AND LOCATIONS:
Overall Officials: Frances Wood, MD, Principal Investigator — WakeMed Health and Hospitals
Locations (1):
- WakeMed, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided